CLINICAL TRIAL: NCT00822068
Title: Improvement of Aphasia After Stroke by Intensive Training and Transcranial Direct Current Stimulation
Brief Title: Improvement of Language Disturbances After Stroke by Intensive Training and Electrical Brain Stimulation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Department of Neurology, University of Muenster
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Aphasia_tDCS
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Aphasia; Stroke
Keywords: stroke; aphasia; rehabilitation; transcranial direct current stimulation; intensive training; chronic aphasia after stroke
MeSH Terms: conditions — Aphasia; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- anodal tDCS (Experimental)
  Interventions: Device: anodal tDCS
- 2 (Active Comparator): cathodal tDCS
  Interventions: Device: cathodal tDCS
- 3 (Placebo Comparator): sham stimulation
  Interventions: Device: sham stimulation

INTERVENTIONS:
Device: anodal tDCS — anodal transcranial direct current stimulation
  Arms: anodal tDCS
Device: cathodal tDCS — cathodal transcranial direct current stimulation
  Arms: 2
Device: sham stimulation — sham stimulation
  Arms: 3

SUMMARY:
The study aims to identify if intensive language training, consisting mainly of computer-based object naming, together with electrical brain stimulation, will lead to an improvement of language functions in patients that suffer from language disturbances after a stroke.

ELIGIBILITY:
Inclusion Criteria:

* chronic stroke (> 1 year after event)
* aphasia due to stroke with naming impairment
* German as first language
* first-ever stroke

Exclusion Criteria:

* more than 1 stroke
* progressive stroke
* history of severe alcohol or drug abuse, psychiatric illnessess like severe depression, poor motivational capacity
* dementia
* contraindications for Magnetic Resonance Imaging

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Number of words correctly named after training plus tDCS | 1 year

SECONDARY OUTCOMES:
Communicative-Activity-Log & Stroke-and-Aphasia-Quality-of-Life-Scale | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Floel, MD, Principal Investigator — Department of Neurology, University of Muenster; Department of Neurology, University of Berlin, Germany
Locations (1):
- Department of Neurology, University of Muenster; Department of Neurology, University of Berlin, Muenster / Berlin, NRW/Berlin-Brandenburg, Germany

REFERENCES:
- [Derived] Floel A, Meinzer M, Kirstein R, Nijhof S, Deppe M, Knecht S, Breitenstein C. Short-term anomia training and electrical brain stimulation. Stroke. 2011 Jul;42(7):2065-7. doi: 10.1161/STROKEAHA.110.609032. Epub 2011 Jun 2. PMID 21636820